CLINICAL TRIAL: NCT06062810
Title: Explore the Relationship Between Single Nucleotide Polymorphisms and Raloxifene Response and Toxicity in Patients With Breast Cancer LCIS
Brief Title: Pharmacogenomics ANDA SNP Clinical Study - Raloxifene and Single Nucleotide Polymorphisms
Acronym: Drugs-SNPs
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, Medical Monitor, Safety Officer, IORG Director, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: ANDA 220176; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); IRB00009424 (Registry Identifier: HHS, IRB); IORG0007849 (Registry Identifier: HHS, IORG); NPI - 1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI - 1023387701 (Registry Identifier: HHS, Health Care Provider Organization); ANDA 220176 (Registry Identifier: FDA, ANDA)
Record Dates: First submitted 2023-09-09; First posted 2023-10-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: LCIS; ER; UGT; SNP; Pharmacogenomics; Gene; Genetics
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: * The usual approach group (Generic-1)
  * The study approach group (Generic-2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No-placebo and random and double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Raloxifene - Usual (Experimental): * Generic-1 - Raloxifene
  * Chemotherapy
  * Generic-1 - raloxifene hydrochloride tablet
  * Raloxifene 60 mg taken orally daily
  * Usual Approach Group (Generic-1)
  Interventions: Drug: Raloxifene - Usual
- Raloxifene - Study (Experimental): * Generic-2 - Raloxifene
  * Chemotherapy
  * Generic-2 - Raloxifene tablet
  * Raloxifene 60 mg taken orally daily
  * Usual Approach Group (Generic-2)
  Interventions: Drug: Raloxifene - Study

INTERVENTIONS:
Drug: Raloxifene - Usual — * Generic-1 - raloxifene hydrochloride tablet
  * Raloxifene 60 mg taken orally daily
  Other Names: Raloxifene Chemotherapy (Generic-1)
  Arms: Raloxifene - Usual
Drug: Raloxifene - Study — * Generic-2 - Raloxifene tablet
  * Raloxifene 60 mg taken orally daily
  Other Names: Raloxifene Chemotherapy (Generic-2)
  Arms: Raloxifene - Study

SUMMARY:
Explore the relationship between drug target ER gene single nucleotide polymorphisms and Raloxifene therapeutic effects in patients with Breast Cancer LCIS, based on Oxford precisely sequencing drug targets' genes.

Explore the relationship between drug target UGT gene single nucleotide polymorphisms and Raloxifene side-effects in patients with Breast Cancer LCIS, based on Oxford precisely sequencing drug targets' genes.

DETAILED DESCRIPTION:
The usual approach group, after breast tissue biopsy, 300 double blind random group separated BC-LCIS patients currently used the Chemotherapy on Generic-1 - raloxifene hydrochloride tablet, 60 mg daily, it will try to look for the relationship between the Raloxifene therapeutic efficacy and the ER SNP Genotyping, after blood draw, to look for the relationship between the Raloxifene therapeutic safety and the UGT SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

The study approach group, after breast tissue biopsy, 300 double blind random group separated BC-LCIS patients currently used the Chemotherapy on Generic-2 - Raloxifene tablet, 60 mg daily, it will try to look for the relationship between the Raloxifene therapeutic efficacy and the ER SNP Genotyping, after blood draw, to look for the relationship between the Raloxifene therapeutic safety and the UGT SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

1. Detect drug target whole gene precision sequence of everyone patient for all 600 recruited double-blind BC-LCIS patients.
2. Mutually compare everyone patient drug target whole gene precision sequence for a total of 600 recruited double-blind BC-LCIS patients.
3. Calculate drug target gene SNPs in all 600 recruited double-blind BC-LCIS patients.
4. Correlate everyone patient drug target gene SNP to everyone patient drug efficacy.
5. Correlate everyone patient drug target gene SNP to everyone patient drug safety.
6. Mutually compare the usual approach group SNPs (300 double blind random group separated BC-LCIS patients) with the study approach group SNPs (300 double blind random group separated BC-LCIS patients).
7. Confirm the relationship between drug target gene SNPs and drug efficacy.
8. Confirm the relationship between drug target gene SNPs and drug safety.

ELIGIBILITY:
* Select 600 Breast Cancer LCIS Patients who are suitable for breast tissue biopsy
* High risk of breast cancer is defined as at least one breast biopsy showing lobular carcinoma in situ (LCIS)
* Dosage Duration at least 90 days
* The usual approach group - Recruit 300 double blind random group separated BC-LCIS patients currently used the Chemotherapy Dose on Generic-1 - raloxifene hydrochloride tablet, after breast tissue biopsy, and, after blood draw, like as the usual approach group.
* The study approach group - Recruit 300 double blind random group separated BC-LCIS patients currently used the Chemotherapy Dose on Generic-2 - raloxifene tablet, after breast tissue biopsy, and, after blood draw, like as the study approach group.

Inclusion Criteria:

1. Clinical diagnosis of Breast Cancer LCIS
2. Clinical breast tissue biopsy diagnosis showing lobular carcinoma in situ (LCIS)
3. Suitable for enough breast tissue biopsy of Breast Cancer LCIS
4. Random and double blind
5. Measurable disease
6. Adequate organ functions
7. Adequate performance status
8. Age 22 years old and over
9. Sign an informed consent form
10. Receive blood-drawing

Exclusion Criteria:

1. Mastectomy
2. Treatment with other anti-cancer therapies and cannot be stopped currently
3. Pregnancy
4. Breast-feeding
5. The patients with other serious intercurrent illness or infectious diseases
6. Have more than one different kind of cancer at the same time
7. Serious Allergy to Drugs
8. Thrombus or Bleed Tendency
9. Serious Risks or Serious Adverse Events of the drug product
10. The prohibition of drug products
11. Have no therapeutic effects
12. Follow up to the most current label

Ages: 24 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postmenopausal Women
Enrollment: 600 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Measure and Report Raloxifene oncology drug target ER SNP Genotypes which are effectiveness associated. | Up to 12 weeks
  * Recruit 300 double blind random group separated Breast Cancer LCIS patients currently using the Chemotherapy dose on Generic-1 - raloxifene (60mg orally daily), after breast tissue biopsy, to be the usual approach group.
  * Recruit 300 double blind random group separated Breast Cancer LCIS patients currently using the Chemotherapy dose on Generic-2 - raloxifene (60mg orally daily), after breast tissue biopsy, to be the study approach group.
  * Measure above every BC-LCIS patient specific Raloxifene oncology drug target ER SNP genotype in Breast Cancer cell whole genome DNA with Oxford precisely sequencing.
  * Report every BC-LCIS patient specific ER SNP genotype in whole genome DNA sequence.
Measure and Report Raloxifene oncology drug target UGT SNP Genotypes which are risk associated. | Up to 12 weeks
  * Recruit 300 double blind random group separated Breast Cancer LCIS patients currently using the Chemotherapy dose on Generic-1 - raloxifene (60mg orally daily), after blood draw, to be the usual approach group.
  * Recruit 300 double blind random group separated Breast Cancer LCIS patients currently using the Chemotherapy dose on Generic-2 - raloxifene (60mg orally daily), after blood draw, to be the study approach group.
  * Measure above every BC-LCIS patient specific Raloxifene oncology drug target UGT SNP genotype in WBC cell whole genome DNA with Oxford precisely sequencing.
  * Report every BC-LCIS patient specific UGT SNP genotype in whole genome DNA sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Han Xu, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. - IORG0007849 - NPI 1023387701; Han Xu, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. - IORG0007849 - NPI 1023387701; Han Xu, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. - IORG0007849 - NPI 1023387701
Locations (1):
- Medicine Invention Design, Inc. - IORG0007849 - NPI 1023387701, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FWA < 00015357 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IRB < 00009424 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search
- See also: IORG < 0007849 > < Medicine Invention Design Incorporation (MIDI) > — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT06062810/Prot_003.pdf
  • Statistical Analysis Plan (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT06062810/SAP_004.pdf
  • Informed Consent Form (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT06062810/ICF_006.pdf